CLINICAL TRIAL: NCT02080533
Title: Feasibility of Slow-paced Respiration Therapy for Treatment of a Symptom Cluster in Pulmonary Arterial Hypertension
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Penn-SON
Record Dates: First submitted 2014-02-20; First posted 2014-03-06 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: pulmonary arterial hypertension; symptoms; dyspnea; fatigue; sleep
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Dyspnea; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single (Experimental): Slow-paced respiration therapy
  Interventions: Other: Slow-paced respiration therapy

INTERVENTIONS:
Other: Slow-paced respiration therapy — The FDA-approved RESPeRATE device contains headphones and a sensor that attaches to the chest to detect inhalation and exhalation. Musical tones synchronize with the respiratory cycle to slowly guide the user to decrease respirations.

SUMMARY:
Pulmonary arterial hypertension (PAH) is a chronic illness characterized by increased pulmonary pressures resulting in right heart failure and premature death. Common symptoms that impair quality of life and functioning are dyspnea, fatigue and sleep disturbance. This trio of symptoms is highly prevalent and forms a symptom cluster (2 or more symptoms that co-occur) in PAH. From a biological, proinflammatory cytokines are implicated in dyspnea, fatigue and sleep disturbance; there is activation of the sympathetic nervous system (SNS) and an inherent inflammatory process in PAH that contributes to the pathophysiology, but the link to this symptom cluster has not been investigated. One novel, treatment for symptom clusters is slow-paced respiration therapy using the FDA-approved device, RESPeRATE. The device contains headphones and a sensor that attaches to the chest to detect inhalation and exhalation. Musical tones synchronize with the respiratory cycle to slowly guide the user to decrease respirations. RESPeRATE moderates effects of the SNS; lowers blood pressure; improves functional capacity and ejection fraction; and significantly decreases pulmonary pressures in left heart failure. The investigators will enroll 10 women with PAH to use the RESPeRATE device to perform slow-paced respiration for 15 minutes per day for 8 weeks to determine the feasibility and effects on the SNS and inflammatory activity and the symptom cluster. The investigator's overall hypothesis is that, as compared to baseline, after eight weeks of therapy women with PAH who receive slow-based respiration therapy will have lower SNS activity and inflammatory levels, and improved dyspnea, fatigue and sleep disturbance.

ELIGIBILITY:
Inclusion Criteria:

* Previous documentation of mean pulmonary artery pressure > 25 mm Hg with a pulmonary capillary wedge pressure (or left ventricular end-diastolic pressure) < 16 mm Hg and PVR > 3 WU at any time before study entry.
* Women with WHO Group I PAH (idiopathic, heritable, or associated with connective tissue disease, congenital heart disease, anorexigens or HIV)
* Targeted PAH therapy at stable dose for 3 months
* Age >21 years
* Ability to perform six minute walk testing without limitations in musculoskeletal function or coordination.
* Informed consent

Exclusion Criteria:

* Age < 21
* Hypotension (blood pressure < 90/60 mmHg)
* Pregnancy
* Chronic Fatigue Syndrome (current or history of)
* Known sleep disorder (obstructive sleep apnea, restless leg syndrome, narcolepsy, current or history of)
* Hospitalized or acutely ill
* Major Depression (current or history of)
* Lung transplant recipient

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-02; Primary Completion 2015-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Adherence to slow-paced respiration therapy. | 10 weeks
  Adherence rates will be assessed by the frequency of days used.

SECONDARY OUTCOMES:
Change in baseline and Week 10 dyspnea scores on the Multidimensional Dyspnea Profile | Baseline and 10 weeks
Change in baseline and Week 10 fatigue scores on the Multidimensional Fatigue Inventory | Baseline and 10 weeks
Change in baseline and Week 10 sleep scores on the Pittsburgh Sleep Quality Index | Baseline and 10 weeks
Change in baseline and Week 10 norepinephrine levels | Baseline and 10 weeks
Change in baseline and Week 10 interleukin-6 levels | Baseline and 10 weeks
Change in baseline and Week 10 tumor necrosis factor-alpha levels | Baseline and 10 weeks
Change in baseline and Week 10 six minute walk test | Baseline and 10 weeks
Change in baseline and Week 10 right ventricular systolic pressure | Baseline and 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lea Ann Matura, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States